CLINICAL TRIAL: NCT07123610
Title: The Relationship Between Mediterranean Diet Education Given to Shift-Working Nurses and Sleep Quality, Physical Activity Level, Blood Parameters, and Anthropometric Measurements
Brief Title: Mediterranean Diet Education in Shift Nurses: Effects on Sleep, Activity, and Health Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Ilayda Ozturk Altuncevahir, Assist. Prof., Bahçeşehir University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: E-85646034-604.01-81176
Record Dates: First submitted 2025-07-31; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Cardiovascular Diseases; Obesity Prevention; Atheroscleroses; Hypertension; Type 2 Diabetes Mellitus (T2DM); Occupational Health; Metabolic Syndrome
Keywords: Nutritional intervention; Circadian rhythm; Metabolic health; Lifestyle modification; Workplace wellness
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Hypertension; Diabetes Mellitus, Type 2; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Shift working nurses (Experimental)
  Interventions: Behavioral: Mediterranean Diet Education Program

INTERVENTIONS:
Behavioral: Mediterranean Diet Education Program — The intervention consists of a 4-week Mediterranean Diet Education Program designed specifically for nurses working rotating shifts.
  The program included four weekly group sessions, each lasting approximately 60 minutes, delivered in-person by a registered dietitian with training in behavioral change and clinical nutrition. Sessions are interactive and supported by visual and printed educational materials.
  Participants receive a printed handbook including a food pyramid graphic, portion guides, weekly shopping lists, and sample menus tailored to shift work schedules. They also gain access to a moderated online discussion group and receive weekly motivational text messages to reinforce key messages.
  No food is provided directly.

SUMMARY:
This study aimed to evaluate the effects of Mediterranean diet education on sleep quality, physical activity levels, blood parameters, and anthropometric measurements among shift-working nurses.

Primary outcomes: Change in Mediterranean diet adherence and sleep quality scores from baseline to post-intervention.

Secondary outcomes: Changes in physical activity levels, anthropometric indices (e.g., BMI, waist-to-hip ratio), and blood parameters (fasting glucose, insulin, HOMA-IR, lipid profile).

DETAILED DESCRIPTION:
Background Shift work misaligns endogenous circadian rhythms with environmental light-dark cycles, predisposing workers to poor sleep, metabolic dysregulation, weight gain and cardiometabolic disease. Observational and experimental evidence indicates that dietary patterns rich in plant foods, monounsaturated fats and lean proteins-exemplified by the Mediterranean diet (MedDiet)-can attenuate inflammation, improve lipid and glycaemic profiles, and enhance subjective well-being. Educational interventions that reinforce MedDiet principles may therefore represent a pragmatic, low-risk strategy to mitigate health risks in shift-working nurses.

Study Desing Design: Single-group, pre-post intervention study Setting: Private general hospital in Muğla, Türkiye Sample Size: 130 nurses (≈80 % women) employed in rotating shifts, aged 18-55 y Allocation: Not applicable (no comparison arm)

Participant Eligibility Inclusion Criteria Registered nurse working ≥3 rotating shifts per month at the study hospital Age 18-55 years Written informed consent Exclusion Criteria Pregnancy or lactation Current participation in another lifestyle or drug trial Diagnosed sleep disorder requiring pharmacotherapy Medical condition necessitating therapeutic diet incompatible with MedDiet principles Inability to attend ≥75 % of education sessions

Intervention Mediterranean Diet Education Programme (Weeks 1-4) Format: Four weekly face-to-face group sessions (60 min each) delivered by a registered dietitian trained in behavioural counselling.

Content:

Session 1: MedDiet pyramid, portion guidance, meal timing for shift workers Session 2: Practical meal planning; reading food labels; healthy cafeteria choices Session 3: Strategies to increase fruit, vegetable, legume and whole-grain intake; recipe demonstrations Session 4: Reducing ultra-processed foods, sugar-sweetened beverages and saturated fats; sustaining behaviour change Materials: Printed handbook (pyramid graphic, shopping lists, sample menus), online discussion forum and weekly motivational text messages.

Fidelity: Sessions follow a standardised script; attendance recorded; 10 % of sessions audited by a second dietitian.

Participants receive no meal provision; they are encouraged to apply learned principles during all shifts. No changes are made to hospital food service.

Data Collection and Management Questionnaires are administered electronically via a secure, password-protected platform. Anthropometric measurements are performed in duplicate by trained research staff following WHO protocols. Blood draws coincide with routine occupational health surveillance to minimise burden and cost. Data are de-identified upon entry; only the principal investigator retains the re-identification key in an encrypted file.

Data analysis The analysis of the data collected in the study was performed using the SPSS 21.0 software. Descriptive statistics such as arithmetic mean, frequency, standard deviation, and percentage values were utilized in the analysis. To determine whether the data showed a normal distribution, skewness and kurtosis values were examined, and these values were found to be between -2 and +2, indicating that the data followed a normal distribution. Accordingly, parametric tests were used for comparisons between groups based on demographic information and for examining relationships between scales. To compare the pre- and post-test results of the Mediterranean diet, sleep disorders, and physical activity scales with blood parameters, the Paired-Samples T-Test was used, while comparisons by gender were conducted using the Independent-Samples T-Test. For comparisons across age groups, One-Way ANOVA was performed, and Tukey's test was applied as the post hoc analysis. Additionally, Pearson correlation analysis was conducted to determine the relationships between nurses' Mediterranean diet education and their sleep quality, physical activity levels, blood parameters, and anthropometric measurements.

The internal consistency of the Mediterranean Diet Adherence Scale, developed by Özkan Pehlivanoğlu, Hüseyin Balcıoğlu, and İlhami Ünlüoğlu, was calculated as Cronbach's α = 0.829, indicating a high level of reliability. The Pittsburgh Sleep Quality Index, developed by Buysse et al. in 1989, demonstrated satisfactory internal consistency (Cronbach's α = 0.80), test-retest reliability, and construct validity. In their 2017 systematic review of physical activity assessment in amputees, Piazza, Ferreira, Minsky, Pires, and Silva reported a reproducibility coefficient of ρ = 0.81 (95% CI = 0.79-0.82).

Outcome Measures and Time Points Primary and secondary outcomes were assessed at baseline (Week 0) and after the intervention (Week 8), unless otherwise specified.

The primary outcomes of the study were adherence to the Mediterranean diet and sleep quality. Adherence was measured using the 14-item Mediterranean Diet Adherence Screener (MEDAS), a validated tool for assessing compliance with Mediterranean dietary principles. Sleep quality was evaluated using the Pittsburgh Sleep Quality Index (PSQI), a widely used self-report instrument for assessing subjective sleep patterns and disturbances.

The secondary outcomes included physical activity level, anthropometric measurements, blood biomarkers, and adverse events. Physical activity was assessed using the International Physical Activity Questionnaire-Short Form (IPAQ-SF). Anthropometric data were collected through standardized procedures: height was measured at baseline using a stadiometer, and weight, body fat percentage, and skeletal muscle mass were evaluated at both time points using the Tanita MC-180 body composition analyzer. Waist and hip circumferences were measured with a non-elastic measuring tape.

Blood biomarkers were assessed via fasting venous blood samples collected and analyzed in the hospital laboratory. Parameters included fasting glucose, insulin, triglycerides, LDL cholesterol, HDL cholesterol, and total cholesterol. The Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) was calculated using fasting glucose and insulin values.

In addition, potential adverse events were monitored continuously throughout the study using a structured questionnaire administered at regular intervals.

Ethical Considerations Ethical approval was obtained from the Bahçeşehir University Scientific Research and Publication Ethics Committee. The study complies with the Declaration of Helsinki and relevant local regulations. Participation is voluntary; nurses may withdraw at any time without affecting employment status or access to occupational health services. The intervention poses minimal risk (education only).

Recruitment begun May 2024 and finished November 2024.

ELIGIBILITY:
Inclusion Criteria:

* Registered nurse working ≥3 rotating shifts per month at the study hospital
* Age 18-55 years
* Written informed consent

Exclusion Criteria:

* Pregnancy or lactation
* Current participation in another lifestyle or drug trial
* Diagnosed sleep disorder requiring pharmacotherapy
* Medical condition necessitating therapeutic diet incompatible with MedDiet principles
* Inability to attend ≥75 % of education session

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2024-05-08 (Actual); Primary Completion 2024-11-09 (Actual); Study Completion 2024-11-09 (Actual)

PRIMARY OUTCOMES:
MEDAS Score | Baseline (week 0) and post-intervention (week 8)
  Change in Mediterranean Diet Adherence Score (MEDAS) Change in adherence to the Mediterranean diet as measured by the 14-item Mediterranean Diet Adherence Screener (MEDAS). This validated questionnaire assesses the frequency and quality of consumption of key Mediterranean dietary components. Scores range from 0 to 14, with higher scores indicating greater adherence.

SECONDARY OUTCOMES:
Change in Physical Activity | Baseline (week 0), Postintervention (week 8)
  Change in physical activity level as measured by the International Physical Activity Questionnaire - Short Form (IPAQ-SF). The IPAQ-SF estimates weekly energy expenditure (in MET-minutes/week) across domains such as walking, moderate and vigorous activity.
BMI Change | Baseline (Week 0) and Post-Intervention (Week 8)
  Change in BMI calculated as weight (kg) divided by height squared (m²). Weight measured using the Tanita MC-180 body composition analyzer; height measured at baseline with a stadiometer. Body Mass Index (BMI) will be calculated using weight and height measurements. Weight was measured in kilograms (kg) and height was measured in meters (m). BMI was computed as weight (kg) divided by the square of height (m²) and reported in kg/m² as a single outcome measure.
Sleep Quality | baseline (week 0) postintervention (week 8)
  Change in sleep quality as measured by the Pittsburgh Sleep Quality Index (PSQI). This 19-item self-report tool assesses subjective sleep quality, latency, duration, efficiency, disturbances, and daytime dysfunction. Scores range from 0 to 21; higher scores indicate poorer sleep quality.
Waist Hip Ratio | Baseline (Week 0) and Post-Intervention (Week 8)
  Change in waist-to-hip ratio (WHR), calculated by dividing waist circumference by hip circumference. Measurements obtained using a non-elastic measuring tape according to WHO standards.
Change in Blood Results Profile | Baseline (Week 0) and Post-Intervention (Week 8)
  Change in fasting blood glucose levels, measured via venous blood draw in a hospital laboratory.
  Changes in fasting insulin levels and HOMA-IR (Homeostatic Model Assessment of Insulin Resistance) Changes in serum lipid parameters, including total cholesterol, LDL cholesterol, HDL cholesterol, and triglycerides, measured from fasting venous blood samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Bodrum Acıbadem Hospital, Muğla, Bodrum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical and privacy considerations.

REFERENCES:
- [Background] Sun M, Feng W, Wang F, Li P, Li Z, Li M, Tse G, Vlaanderen J, Vermeulen R, Tse LA. Meta-analysis on shift work and risks of specific obesity types. Obes Rev. 2018 Jan;19(1):28-40. doi: 10.1111/obr.12621. Epub 2017 Oct 4. PMID 28975706
- [Background] Franzago M, Alessandrelli E, Notarangelo S, Stuppia L, Vitacolonna E. Chrono-Nutrition: Circadian Rhythm and Personalized Nutrition. Int J Mol Sci. 2023 Jan 29;24(3):2571. doi: 10.3390/ijms24032571. PMID 36768893